CLINICAL TRIAL: NCT00003913
Title: A Multicenter Study of Unrelated Umbilical Cord Blood as an Alternate Source of Stem Cells for Transplantation
Brief Title: Umbilical Cord Blood Transplantation in Treating Patients With Hematologic Cancer or Nonmalignant Hematologic Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 1330.00; FHCRC-1330.00; UMN-MT-9817; NCI-G99-1523; CDR0000067092 (Registry Identifier: PDQ); NCT00053755 (obsolete NCT alias)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-03

CONDITIONS: Leukemia; Lymphoma; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: recurrent childhood acute lymphoblastic leukemia; recurrent childhood lymphoblastic lymphoma; recurrent childhood acute myeloid leukemia; relapsing chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; childhood acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; recurrent/refractory childhood Hodgkin lymphoma; refractory anemia; refractory anemia with ringed sideroblasts; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; chronic myelomonocytic leukemia; acute undifferentiated leukemia; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; juvenile myelomonocytic leukemia; blastic phase chronic myelogenous leukemia; childhood chronic myelogenous leukemia; atypical chronic myeloid leukemia; myelodysplastic/myeloproliferative disease, unclassifiable
MeSH Terms: conditions — Leukemia; Lymphoma; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Recurrence; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic; Leukemia, Biphenotypic, Acute; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Leukemia, Myelomonocytic, Juvenile; Blast Crisis; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders | interventions — Antilymphocyte Serum; Filgrastim; Busulfan; Cyclophosphamide; Methylprednisolone; Cord Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: anti-thymocyte globulin
Biological: filgrastim
Drug: busulfan
Drug: cyclophosphamide
Drug: methylprednisolone
Procedure: umbilical cord blood transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Umbilical cord blood transplantation may be able to replace immune cells that were destroyed by the chemotherapy or radiation therapy that was used to kill cancer cells.

PURPOSE: Phase II trial to study the effectiveness of umbilical cord blood transplantation plus combination chemotherapy in treating patients who have hematologic cancer or nonmalignant hematologic disease.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of umbilical cord blood transplantation, as measured by durable neutrophil engraftment, in patients with malignant or nonmalignant hematological disease.
* Determine the disease-free survival and long-term survival in patients treated with this regimen.
* Determine the incidence of neutrophil engraftment, primary and secondary graft failure, platelet engraftment, and RBC engraftment in patients treated with this regimen.
* Determine the incidence and severity of acute and chronic graft-versus-host disease, complications (infection, veno-occlusive disease, interstitial pneumonitis), relapse, other malignancies, lymphoproliferative disorders, and posttransplantation myelodysplasia in patients treated with this regimen.
* Determine the immune reconstitution in patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients are stratified according to disease group (malignant vs nonmalignant). Patients with malignant disease are further stratified according to quality of HLA match (1 or 2/6 vs 3/6 vs 4/6 vs 5/6 or 6/6), cell dose, and age.

Patients are assigned to one of three conditioning regimens, depending on disease.

* Group A (malignant disease ): Patients undergo total body irradiation (TBI) once on day -8 and twice daily on days -7 to -4. Male patients with acute lymphocytic leukemia (ALL) undergo radiotherapy boost to testes. Patients receive cyclophosphamide (CTX) IV on days -3 and -2 and methylprednisolone (MePRDL) IV and anti-thymocyte globulin (ATG) IV on days -3 to -1.
* Group B (inborn errors of metabolism/storage disease): Patients receive oral busulfan (BU) every 6 hours on days -6 and -5, CTX IV on days -4 and -3, and MePRDL IV and ATG IV every 12 hours on days -2 and -1.
* Group C (other nonmalignant diseases): Patients receive oral BU every 6 hours on days -9 to -6, CTX IV on days -5 to -2, and MePRDL IV and ATG IV on days -3 to -1.

Patients in all groups receive cord blood IV over a maximum of 30 minutes on day 0. Patients also receive MePRDL IV with the first half of the infusion administered immediately before the cord blood infusion and filgrastim (G-CSF) IV beginning 4 hours after transplantation and continuing until blood counts recover.

Patients are followed at 30, 60, and 90 days; at 6 months; and then annually thereafter.

PROJECTED ACCRUAL: Approximately 390 patients will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following diagnoses:

  * Acute myeloid leukemia (AML), with or without myelodysplastic syndromes

    * Not in first complete remission (CR)* with translocations t(8;21) and inv (16) unless failure of first-line induction therapy
    * Not in first CR* with translocations t(15;17) abnormality unless:

      * Failure of first-line induction therapy OR
      * Molecular evidence of persistent disease
    * Not in first CR with Down syndrome
    * Patients with third or greater medullary relapse or refractory disease (other than primary induction failures) receive busulfan/melphalan conditioning regimen NOTE: * CR defined by no greater than 5% blasts in marrow
  * Acute lymphocytic leukemia (ALL)

    * Not in first CR OR
    * High-risk ALL in first CR, with high risk defined as one of the following:

      * Hypoploidy (no greater than 44 chromosomes)
      * Pseudodiploidy with translocations or molecular evidence of t(9;22), 11q23, or t(8;14) (except B-cell ALL) with or without MLL gene arrangement
      * Elevated WBC at presentation

        * Age 6-12 months: greater than 100,000/mm^3
        * Age 10-17 years: greater than 200,000/mm^3
        * Age 18: greater than 20,000/mm^3
      * Failed to achieve CR after 4 weeks of induction therapy
    * Patients with B-ALL must not be in first CR, must meet at least one of the high-risk criteria specified above, or must not meet any of the following criteria:

      * Translocation t(8;14)
      * Blasts have surface immunoglobulins
      * CD10 positive
    * Patients with third or greater medullary relapse or refractory disease (other than primary induction failures) receive busulfan/melphalan conditioning regimen
  * Chronic myelogenous leukemia, meeting criteria for 1 of the following:

    * Accelerated phase
    * Chronic phase if 1 year from diagnosis without a matched unrelated bone marrow donor AND unresponsive to or unable to tolerate interferon
    * Blast crisis, defined as greater than 30% promyelocytes plus blasts in bone marrow

      * Patients receive busulfan/melphalan conditioning regimen
  * Acute undifferentiated leukemia (AUL), infant leukemia, or biphenotypic leukemia

    * Patients with third or greater medullary relapse or refractory disease (other than primary induction failures) receive busulfan/melphalan conditioning regimen
  * Juvenile myelomonocytic leukemia meeting the following criteria:

    * No Philadelphia chromosome
    * Bone marrow blasts less than 30%
    * Peripheral blood monocytes greater than 1,000/mm^3
    * At least 2 of the following:

      * Peripheral blood spontaneous growth and/or sargramostim (GM-CSF) hypersensitivity
      * Increased hemoglobin F for age
      * Clonal abnormalities (e.g., monosomy 7 or RAS mutations)
      * Peripheral blood with myeloid precursors
      * WBC greater than 10,000/mm^3
  * Myelodysplastic syndromes defined by the following:

    * Refractory anemia (RA)
    * RA with ringed sideroblasts
    * RA with excess blasts (RAEB)
    * RAEB in transformation
    * Chronic myelomonocytic leukemia
  * Paroxysmal nocturnal hemoglobinuria
  * Hodgkin's lymphoma or non-Hodgkin's lymphoma beyond first CR or primary induction failures AND chemosensitive (greater than 50% reduction in tumor mass size)
  * Inborn error of metabolism including, but not limited to, Hurler's syndrome, adrenoleukodystrophy (ALD), Maroteaux-Lamy syndrome, globoid cell leukodystrophy, metachromatic leukodystrophy, fucosidosis, or mannosidosis

    * For ALD patients over age 5, IQ must be at least 80
    * For all other patients over age 5, IQ must be at least 70
    * For all patients age 5 and under, developmental quotient or clinical neurodevelopmental examination should demonstrate potential for stabilization at a level of functioning where continuous life support (e.g., mechanical ventilation) would not be predicted to be required in the year after transplantation
  * Combined immune deficiencies including, but not limited to:

    * Severe combined immunodeficiency (SCID) requiring cytoreduction
    * Wiskott-Aldrich syndrome
    * Leukocyte adhesion defect
    * Chediak-Higashi disease
    * X-linked lymphoproliferative disease
    * Adenosine deaminase deficiency
    * Purine nucleoside phosphorylase deficiency
    * X-linked SCID
    * Common variable immune deficiency
    * Nezelof's syndrome
    * Cartilage hair hypoplasia
* No dyskeratosis congenita
* No ALL, AML, AUL, or biphenotypic leukemia in third or higher medullary relapse or refractory disease other than primary induction failure
* No primary myelofibrosis or myelofibrosis grade 3 or worse
* No active CNS leukemia involvement (CSF with WBC greater than 5/mm^3 and malignant cells on cytospin)
* No consenting 5/6 or 6/6 HLA-matched related donor available
* 3-6/6 HLA-matched unrelated umbilical cord blood donor available

PATIENT CHARACTERISTICS:

Age:

* See Disease Characteristics
* 18 and under

Performance status:

* Karnofsky 70-100%, if age 16 to 18
* Lansky 50-100%, if under age 16

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Bilirubin less than 2.5 mg/dL
* SGOT less than 5 times upper limit of normal

Renal:

* Creatinine normal for age OR
* Creatinine clearance or glomerular filtration rate greater than 50% lower limit of normal for age

Cardiovascular:

* If symptomatic:

  * LVEF greater than 40% (or shortening fraction greater than 26%) and improves with exercise OR
  * Shortening fraction greater than 26%

Pulmonary:

* If symptomatic:

  * DLCO, FEV_1, and FEC greater than 45% predicted OR
  * Oxygen saturation greater than 85% on room air

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No uncontrolled viral, bacterial, or fungal infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* At least 1 year since prior allogeneic stem cell transplantation (SCT) with cytoreductive preparative therapy
* At least 6 months since prior autologous SCT
* No concurrent thrombopoietic growth factors

Chemotherapy:

* See Disease Characteristics
* See Biologic therapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 390 (Estimated)
Dates: Start 1998-12; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Delaney, MD, MSC, Study Chair — Fred Hutchinson Cancer Center
Locations (23):
- United States (23):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Warren Grant Magnuson Clinical Center, Bethesda, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Spectrum Health and DeVos Children's Hospital, Grand Rapids, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - North Shore University Hospital, Manhasset, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical City Dallas Hospital, Dallas, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington